CLINICAL TRIAL: NCT04541875
Title: A Longitudinal, Digital Study Using the Medication Adherence Reasons Scale (MAR-Scale) to Identify the Reasons for Non-adherence to Medications in Rare Disease
Brief Title: Medication Adherence and Non-adherence in Adults With Rare Disease
Status: Withdrawn | Type: Observational
Why Stopped: Liquidation of sponsor
Sponsor: Xperiome (Other)
Collaborators: The Touro College and University System (Other)
Responsible Party: Sponsor
Other Study IDs: RM-RP005
Record Dates: First submitted 2020-08-26; First posted 2020-09-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Cystic Fibrosis; Hemophilia A; Hemophilia B; Idiopathic Pulmonary Fibrosis; Myasthenia Gravis; Sickle Cell Disease
Keywords: Adherence; MAR-Scale; Rare disease; Observational
MeSH Terms: conditions — Cystic Fibrosis; Hemophilia A; Hemophilia B; Idiopathic Pulmonary Fibrosis; Myasthenia Gravis; Anemia, Sickle Cell; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cystic fibrosis: Patients aged 18+ and diagnosed with cystic fibrosis.
  Patients will answer the MAR-Scale once every three months for a year.
  Interventions: Other: MAR-Scale
- Hemophilia A or B: Patients aged 18+ and diagnosed with hemophilia A or B.
  Patients will answer the MAR-Scale once every three months for a year.
  Interventions: Other: MAR-Scale
- Idiopathic pulmonary fibrosis: Patients aged 18+ and diagnosed with idiopathic pulmonary fibrosis.
  Patients will answer the MAR-Scale once every three months for a year.
  Interventions: Other: MAR-Scale
- Myasthenia gravis: Patients aged 18+ and diagnosed with myasthenia gravis.
  Patients will answer the MAR-Scale once every three months for a year.
  Interventions: Other: MAR-Scale
- Sickle cell disease: Patients aged 18+ and diagnosed with sickle cell disease.
  Patients will answer the MAR-Scale once every three months for a year.
  Interventions: Other: MAR-Scale

INTERVENTIONS:
Other: MAR-Scale — The MAR-Scale is a 20-item questionnaire based on commonly reported reasons for non-adherence to medications.

SUMMARY:
The purpose of this study is to use the Medication Adherence Reasons Scale (MAR-Scale) to determine the extent of non-adherence to specific medications indicated to treat cystic fibrosis, hemophilia (A or B), idiopathic pulmonary fibrosis, myasthenia gravis, and sickle cell disease, and to identify the top patient-reported reasons for non-adherence. Internal reliability of the MAR-Scale will also be assessed in each condition.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed (self-reported) diagnosis by a doctor or other licensed healthcare professional of one of the following conditions:
* Cystic fibrosis
* Hemophilia (A or B)
* Idiopathic pulmonary fibrosis
* Myasthenia gravis
* Sickle cell disease
* Have access to the internet
* Are aged 18 years or above
* Are comfortable reading and answering questions in English
* Have an active prescription for at least one medication indicated to treat the relevant condition (self-reported)
* NB: Individuals will be eligible even if the prescription has not been dispensed (filled) yet, and also if they have the medication(s), but are not actually taking it/them Are able and willing to provide consent electronically through the my.raremark.com platform

Exclusion Criteria:

* There are no exclusion criteria. Any member of a Raremark community will be able to take part in this study if they meet the inclusion criteria and can provide their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone who fits the eligibility criteria and gives their consent to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
To use the MAR-Scale to determine the extent of non-adherence to specific medications indicated to treat a range of rare diseases. | Baseline
  Percentage of respondents who indicated at least one reason for non-adherence in the past seven days.
To use the MAR-Scale to determine the extent of non-adherence to specific medications indicated to treat a range of rare diseases. | 3 months
  Percentage of respondents who indicated at least one reason for non-adherence in the past seven days.
To use the MAR-Scale to determine the extent of non-adherence to specific medications indicated to treat a range of rare diseases. | 6 months
  Percentage of respondents who indicated at least one reason for non-adherence in the past seven days.
To use the MAR-Scale to determine the extent of non-adherence to specific medications indicated to treat a range of rare diseases. | 9 months
  Percentage of respondents who indicated at least one reason for non-adherence in the past seven days.
To use the MAR-Scale to determine the extent of non-adherence to specific medications indicated to treat a range of rare diseases. | 1 year
  Percentage of respondents who indicated at least one reason for non-adherence in the past seven days.
To use the MAR-Scale to identify the top patient-reported reasons for non-adherence to specific medications indicated to treat these rare diseases. | Baseline
  Tally of reasons for non-adherence.
To use the MAR-Scale to identify the top patient-reported reasons for non-adherence to specific medications indicated to treat these rare diseases. | 3 months
  Tally of reasons for non-adherence.
To use the MAR-Scale to identify the top patient-reported reasons for non-adherence to specific medications indicated to treat these rare diseases. | 6 months
  Tally of reasons for non-adherence.
To use the MAR-Scale to identify the top patient-reported reasons for non-adherence to specific medications indicated to treat these rare diseases. | 9 months
  Tally of reasons for non-adherence.
To use the MAR-Scale to identify the top patient-reported reasons for non-adherence to specific medications indicated to treat these rare diseases. | 1 year
  Tally of reasons for non-adherence.

SECONDARY OUTCOMES:
To perform psychometric analysis of the MAR-Scale questionnaire based on data collected from rare disease patients. | Baseline
  Use the 200 responses collected from each condition to determine the Cronbach's alpha of the scale for each condition.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Unni, BpharmMBAPhD, Principal Investigator — Touro College of Pharmacy

IPD SHARING:
Plan to Share IPD: Undecided